CLINICAL TRIAL: NCT07058480
Title: Combined Muscle Energy Technique and Myofascial Chain Stabilization Reduces Menstrual Pain and Improves Pelvic Alignment in Women With Primary Dysmenorrhea: A Prospective Study
Brief Title: Muscle Energy Technique and Myofascial Chain Training for Menstrual Pain in Primary Dysmenorrhea (METPD-25)
Acronym: METPD-25
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanjiao Luo (Other)
Responsible Party: Sponsor-Investigator, Shanjiao Luo, PhD Candidate / Principal Investigator, Shenzhen Jianan Hospital
Organization: Shenzhen Jianan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JAH-METPD-2025-01
Record Dates: First submitted 2025-06-23; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Primary Dysmenorrhea (PD)
Keywords: Pelvic Girdle Dysfunction; Muscle Energy Technique; Pelvic Stabilization Training; Pelvic Alignment
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: This study adopted a prospective, two-arm parallel assignment design to compare the effects of MET combined with myofascial chain-based pelvic stabilization training versus conventional physiotherapy in women with primary dysmenorrhea.
Masking Description: This was an open-label study without any masked parties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined MET and MFC-Based Pelvic Stabilization (Experimental): Participants receive Muscle Energy Technique (MET) for iliac dysfunction and sacral torsion, plus myofascial chain-based pelvic stabilization training (curl-ups, planks, anti-rotation). 3 sessions/week, 50 minutes/session, for 4 weeks.
  Interventions: Behavioral: Combined MET and MFC-Based Pelvic Stabilization Training
- Interferential current therapy (ICT) and Deep Friction Massage (DFM) (Active Comparator): Participants receive medium- and low-frequency electrotherapy and deep friction massage targeting the lumbar (lower back), sacroiliac, and iliac crest regions. 3 sessions/week, 50 minutes/session, for 4 weeks.
  Interventions: Device: Interferential current therapy (ICT); Behavioral: Deep Friction Massage (DFM)

INTERVENTIONS:
Behavioral: Combined MET and MFC-Based Pelvic Stabilization Training — This intervention consisted of a combination of Muscle Energy Technique (MET) for iliac and sacral dysfunctions (20 minutes per session) and myofascial chain-based pelvic stabilization training (including curl-ups, planks, and anti-rotation exercises; 30 minutes per session), targeting pelvic alignment and neuromuscular control. Sessions were conducted 3 times per week, 50 minutes per session, for 4 consecutive weeks.
  Arms: Combined MET and MFC-Based Pelvic Stabilization
Device: Interferential current therapy (ICT) — Interferential current therapy (ICT) was applied to the lumbar (lower back), sacroiliac, and iliac crest regions, 3 sessions per week, 20 minutes per session, for 4 weeks.
  Arms: Interferential current therapy (ICT) and Deep Friction Massage (DFM)
Behavioral: Deep Friction Massage (DFM) — Deep friction massage was administered to the lumbar, sacroiliac, and iliac crest regions for 30 minutes per session, 3 sessions per week, for 4 weeks.
  Arms: Interferential current therapy (ICT) and Deep Friction Massage (DFM)

SUMMARY:
This prospective clinical trial evaluates the effects of a non-pharmacological intervention combining muscle energy technique (MET) and myofascial chain (MFC)-based pelvic stabilization training in women with primary dysmenorrhea (PD). The study aims to determine whether this combined approach can improve pelvic alignment, reduce menstrual pain, and enhance static balance. Participants are assigned to either an experimental group receiving MET + MFC-based training or a control group receiving conventional physiotherapy. Outcomes include radiographic pelvic parameters, pain intensity, and balance performance.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is a common gynecological condition characterized by cyclic lower abdominal pain without an identifiable organic cause. Biomechanical factors such as pelvic misalignment and myofascial imbalance are increasingly recognized as contributing to the persistence and severity of PD.

This prospective non-randomized controlled trial investigates whether a combined intervention of muscle energy technique (MET) and myofascial chain (MFC)-based pelvic stabilization training can improve pelvic structure and reduce clinical symptoms in women with PD. Participants are women aged 18-45 years with moderate-to-severe PD and radiographic evidence of pelvic misalignment. They are assigned to one of two groups:

Experimental group: MET plus MFC-based core stabilization exercises. Control group: Interferential current therapy and deep friction massage. Interventions are administered three times per week for four weeks. The primary outcomes include changes in pelvic sagittal parameters (pelvic tilt, sacral slope, pelvic incidence), pelvic symmetry, menstrual pain (measured by VAS), and static balance (eyes-closed single-leg stance). Assessments are conducted at baseline, 4 weeks, and 12 weeks post-intervention.

The study aims to explore whether biomechanical correction of pelvic alignment contributes to pain modulation and functional improvement in women with PD, providing a basis for non-pharmacological rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-45 years
* Regular menstrual cycles
* Clinically diagnosed with primary dysmenorrhea
* Visual Analog Scale (VAS) score ≥ 4 during menstruation for at least six consecutive months
* Radiographic evidence of pelvic tilt, sacral slope deviation, or frontal pelvic asymmetry

Exclusion Criteria:

* Secondary dysmenorrhea or diagnosed gynecological pathologies (e.g., endometriosis, ovarian cysts)
* Pregnancy or lactation
* Current use of hormonal contraceptives or hormone therapy
* Ongoing or recent physical therapy targeting the pelvis
* History of pelvic or spinal surgery
* Congenital or structural musculoskeletal disorders affecting the lumbopelvic region

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study specifically targets biologically female participants of reproductive age who experience moderate to severe primary dysmenorrhea, as defined by VAS ≥ 4.
Enrollment: 30 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change in menstrual pain intensity measured by Visual Analog Scale (VAS) | Baseline (pre-intervention), Week 4 (immediate post-intervention), and Week 12 (telephone follow-up to assess sustainability of treatment effects)
  The primary outcome was the change in pain intensity before and after intervention, assessed using the Visual Analog Scale (VAS，0-10). Participants rated their average menstrual pain during the most painful day of menstruation. A reduction in VAS score indicated improvement in dysmenorrhea symptoms.

SECONDARY OUTCOMES:
Change in Pelvic Tilt (PT) Angle | Baseline and Week 4 (end of intervention)
  Change in PT (degrees) from baseline to Week 4, assessed by standardized lateral pelvic radiograph.
Change in Sacral Slope (SS) Angle | Baseline and Week 4 (end of intervention)
  Change in SS (degrees) from baseline to Week 4, assessed by standardized lateral pelvic radiograph.
Change in Pelvic Incidence (PI) Angle | Baseline and Week 4 (end of intervention)
  Change in PI (degrees) from baseline to Week 4, assessed by standardized lateral pelvic radiograph.
Change in Pelvic Asymmetry Score | Baseline and Week 4 (end of intervention)
  Change in pelvic asymmetry assessed by frontal pelvic X-rays from baseline to Week 4. Pelvic asymmetry is determined by a composite score based on iliac crest height discrepancy, anterior/posterior innominate rotation, adduction/abduction shift, and sacral torsion.
Change in Static Balance | Baseline and Week 4 (end of intervention)
  Change in single-leg stance time (seconds, eyes closed) from baseline to Week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Shanjiao Luo, PhD, Principal Investigator — Shenzhen JianAn Hospital / Sehan University
Locations (1):
- Shenzhen JianAn Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome results reported in the manuscript will be shared. This includes demographic information, baseline measurements, and outcome data at each time point (e.g., VAS, pelvic alignment, and balance test results). No personally identifiable information will be disclosed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documentation will be available from 6 months after publication of the results in a peer-reviewed journal. The data will be accessible for a period of 2 years via request to the corresponding author (luoshanjiao@gmail.com).
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to the de-identified individual participant data (IPD) and supporting documents. Requests should be directed to the corresponding author via email (luoshanjiao@gmail.com). Access will be granted on a case-by-case basis after approval by the study team.
URL: https://clinicaltrials.gov

REFERENCES:
- [Background] Gartenberg A, Nessim A, Cho W. Sacroiliac joint dysfunction: pathophysiology, diagnosis, and treatment. Eur Spine J. 2021 Oct;30(10):2936-2943. doi: 10.1007/s00586-021-06927-9. Epub 2021 Jul 16. PMID 34272605
- [Background] Ju H, Jones M, Mishra G. The prevalence and risk factors of dysmenorrhea. Epidemiol Rev. 2014;36:104-13. doi: 10.1093/epirev/mxt009. Epub 2013 Nov 26. PMID 24284871
- [Background] Wang J, He X, Zhu C, Ding H, Feng G, Yang X, Liu L, Song Y. The relationship between spino-pelvic alignment and primary dysmenorrhea. Front Surg. 2023 Feb 8;10:1125520. doi: 10.3389/fsurg.2023.1125520. eCollection 2023. PMID 36843999
- [Background] Legaye J, Duval-Beaupere G, Hecquet J, Marty C. Pelvic incidence: a fundamental pelvic parameter for three-dimensional regulation of spinal sagittal curves. Eur Spine J. 1998;7(2):99-103. doi: 10.1007/s005860050038. PMID 9629932
- See also: Shenzhen JianAn Hospital official website, the clinical trial site. — http://www.jayy.cn

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT07058480/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT07058480/ICF_001.pdf